CLINICAL TRIAL: NCT03251794
Title: Ultrasonographic Evaluation of Fetal Adrenal Gland in Cases of Threatened Preterm Labor
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: FAGE
Record Dates: First submitted 2017-08-13; First posted 2017-08-16 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- threatened preterm labor: women presented to the reception unit from 28-37 weeks by regular contractions and opened cervix
  Interventions: Diagnostic Test: three dimensional ultrasound; Diagnostic Test: color Doppler

INTERVENTIONS:
Diagnostic Test: three dimensional ultrasound — evaluation of the suprarenal glands
Diagnostic Test: color Doppler — Doppler evaluation of the suprarenal artery

SUMMARY:
Preterm birth continues to be a major public health problem with lasting family and societal repercussions. Despite tremendous research effort, prevention strategies have failed, and the prevalence of preterm birth in the United States reached 12.3% in 2003.

Prematurity causes 70% of fetal/neonatal deaths. 11.4% of births are at < 37 weeks' gestation. The rate of prematurity increases dramatically with the number of fetuses - singletons 10%; twins 54.9%; and triplets 93.6%

ELIGIBILITY:
Inclusion Criteria:

1. singleton fetus less than 37 weeks of gestation
2. women diagnosed to having Threatened preterm labor.

   1. presence of uterine contraction (at least 4 in 20 min or 8 in 60 min )
   2. cervical effacement <80 %
   3. cervical dilatation <1 cm

Exclusion Criteria:

1. suspected fetal growth restriction,
2. maternal medical complications,
3. presence of fetal heart rate abnormalities at enrollment.
4. Preterm Premature rupture of membranes
5. Placenta previa
6. Lower urinary tract infection or genital infection
7. Fetal congenital anomaly

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women with threatened preterm labor
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
the volume of adrenal gland | 5 minutes
  measurement by three dimensional ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided